CLINICAL TRIAL: NCT03440359
Title: "Supplementation of the Luteal Phase With Vaginal Progesterone (Crinone 8%) in Women With Polycystic Ovary Syndrome Undergoing Ovulation Induction With Letrozole: A Prospective and Randomized Controlled Trial
Brief Title: Vaginal Progesterone Supplementation in Women With PCOS Undergoing Ovulation Induction With Letrozole
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Watson Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Laurel Stadtmauer, Principal Investigator, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB 12-07-FB-0170
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS, crinone, vaginal progesterone, ovulation induction
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Crinone; Vaginal Creams, Foams, and Jellies; Letrozole; Ovidrel

STUDY DESIGN:
Intervention Model Description: Participants who met criteria were randomized to either Crinone vaginal therapy versus no therapy in the luteal phase of an ovulation induction cycle. Participants who did not achieve a pregnancy were able to participate in up to 3 cycles, and were re-randomized with each cycle.
Who Masked: Outcomes Assessor
Masking Description: Data analysis was completed by blinded observer who had access only to participant ID number, cycle number and treatment, and pregnancy outcome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- # 1- no progesterone therapy (Other): Letrrozole 2.5 to 5 mg oral tablet cycle day 3-7.Pelvic ultrasound at cycle day 11 or 12 and repeat if needed until leading follicle is >17 mm. Ovidrel 250 mcg injected sq. Timed intercourse or intrauterine insemination. No supplemental progesterone therapy in luteal phase
  Interventions: Drug: Letrozole Oral Tablet; Diagnostic Test: pelvic ultrasound; Drug: Ovidrel 250 MCG Per 0.5 ML Prefilled Syringe; Other: Intrauterine insemination or timed intercourse
- # 2 - Progesterone Vaginal Gel 8% (Active Comparator): Letrrozole 2.5 to 5 mg oral tablet cycle day 3-7. Pelvic ultrasound at cycle day 11 or 12 and repeat if needed until leading follicle is >17 mm. Ovidrel 250 mcg injected sq. Timed intercourse or intrauterine insemination.Crinone 8% (progesterone) vaginal therapy was provided in luteal phase for 14 days .Administration was started the second day after intrauterine insemination or timed intercourse.
  Interventions: Drug: Progesterone Vaginal Gel 8%; Drug: Letrozole Oral Tablet; Diagnostic Test: pelvic ultrasound; Drug: Ovidrel 250 MCG Per 0.5 ML Prefilled Syringe; Other: Intrauterine insemination or timed intercourse

INTERVENTIONS:
Drug: Progesterone Vaginal Gel 8% — progesterone supplementation for luteal phase support administered with vaginal applicators and used instead of progesterone intramuscular injections or progesterone vaginal suppositories.
  Other Names: Crinone 8% vaginal gel
  Arms: # 2 - Progesterone Vaginal Gel 8%
Drug: Letrozole Oral Tablet — letrozole oral tablet 2.5 mg or 5 mg administered cycle day 3-7 for ovulation induction
Diagnostic Test: pelvic ultrasound — pelvic ultrasound performed at cycle day 11 or 12 and repeated as necessary until leading follicle size is >17 mm in diameter
Drug: Ovidrel 250 MCG Per 0.5 ML Prefilled Syringe — ovidrel 250 mcg given when leading follicle size is > 17 mm in diameter
  Other Names: recombinant hCG 250 mcg
Other: Intrauterine insemination or timed intercourse — Intrauterine insemination or timed intercourse (depending on semen parameters) performed 36-40 hours after Ovidrel

SUMMARY:
Aromatase inhibitors such as letrozole are hypothesized to maintain normal hypothalamic/ pituitary feedback mechanisms and in the case of OI (ovulation induction) in women with PCOS, may act to increase follicular sensitivity to FSH by increasing intrafollicular androgen levels. Letrozole also may act to increase midluteal P levels presumably by induction of follicles and corpora lutea. The investigators are asking the question whether P supplementation with Crinone (8%) may have an additive beneficial effect on endometrial development in those women taking letrozole. Progesterone levels in the endometrium (tissue levels) have been documented to be significantly higher than serum levels after vaginal administration which may lead to higher pregnancy rates. In addition P has been shown to decrease LH pulse frequency which is elevated in PCOS and has been shown to down regulate endometrial androgen receptors. There have been retrospective studies showing progesterone supplementation seems to benefit both CC and letrozole treatment groups. In fact, this study showed the only pregnancies in the letrozole group were those in women who took P supplementation. However the number of cycles studied was small. There is a place for a randomized controlled trial (RCT) to determine if luteal phase P supplementation with Crinone should be used in all women using letrozole for Ovulation Induction (OI) in combination with Intrauterine Insemination (IUI) or Timed Intercourse (TI). This is currently not done in all clinical practices.

DETAILED DESCRIPTION:
Approval of the study was obtained from the local IRB. Prospective volunteers had had an infertility workup including blood hormone levels (FSH, LH, E2, Progesterone, Prolactin, and Thyroid), partner's semen analysis, HSG, laparoscopy or hydrosonogram, plus a baseline evaluation including ultrasound of ovaries and uterus performed as standard of care. If the results of these tests and the remaining Inclusion/Exclusion criteria were met, the study consent was reviewed with participants and signatures were obtained. Participants contacted the clinic at the start of their menses (spontaneous or progesterone-induced) to start the treatment cycle. Eligibility criteria was reviewed, and Letrozole 2.5-7.5 mg day 3-7 was initiated based on BMI and prior response. An ultrasound was performed on cycle day 11 or 12 and repeated if needed to determine response until at least 1 follicle with mean diameter > 17mm in size was observed. When the appropriate follicle size was reached, participants were randomized into one of the two treatment groups as determined by a randomization table, and Ovidrel (250mcg) was administered. If there was no response identified by follicle growth on day 21, the participant was considered a letrozole failure, the cycle was stopped, and the participant was dropped from the study and was not included in subsequent cycles.

IUI/TI was performed at 24-48 hours after the Ovidrel (hCG) injection. If the participant was randomized to progesterone (Crinone), the luteal phase was supplemented once daily with vaginal progesterone (Crinone 8%) starting the second day after the IUI or TI and continued for 14 days. A urine or serum pregnancy test was performed as standard of care 16 days after the IUI/TI. If the test was positive, a confirmatory blood level (βhCG) was performed as standard of care X2 (1 week apart) and an ultrasound on post-hCG day 35-42 was done. Any pregnancies occurring in either treatment group were followed for delivery outcomes. Information regarding the delivery (induced, vaginal, cesarean section), date of birth, infant measurements (weight and length) and other important information regarding the infant's condition was obtained. Participants were allowed to undergo up to 3 cycles of letrozole as the pregnancy rates for the first 3 cycles have been shown to be similar. The participants were re-randomized each cycle. If the participant was pregnant, Crinone (8%) was continued until 10 weeks gestation in both groups.

Each participant was able to proceed with up to 3 cycles (consecutively, if desired) of OI over the next 6 months and was re-randomized each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Women who have anovulatory or oligoovulatory infertility who are undergoing ovulation induction for infertility with TI or IUI , with or without regular cycles defined as cycle length > 35 days, < 26 days or amenorrhea (no cycles in the past six months), and who meet 2 out of 3 of the Rotterdam Criteria (1. Chronic anovulation or irregular cycles, 2. Clinical or biochemical hyperandrogenism, 3. Polycystic appearing ovaries on ultrasound.)
* Day 3 FSH(Follicle stimulating hormone)< 10 (obtained within 2 years prior to screening
* Documented infertility for at least 1 year or documented anovulation
* Willing to participate in up to 3 cycles of OI with letrozole and IUI or TI
* Partner's or donor's SA> 5 million motile sperm within 2 years of screening
* Patients may have received clomiphene citrate or letrozole treatment in the past.

Exclusion Criteria:

* Untreated thyroid or prolactin abnormalities
* Pregnancy in the last 3 months
* BMI< 18 or >40kg/m2
* Abnormal uterine bleeding of undetermined origin
* Contraindications to pregnancy
* Progesterone sensitivity
* Uterine anomalies seen on ultrasound (performed within 6 months prior to screening) that can affect pregnancy chances such as submucosal uterine fibroids or polyps
* Three or more previous consecutive pregnancy losses
* Blocked fallopian tubes X2 (documented by HSG, laparoscopy, or hydrosonogram completed within past 3 years)
* More than 3 failed monitored letrozole cycles prior to enrolling

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates | Per initiated cycle of treatment. At the end of Cycle 1, 2, and 3 (each cycle is 28 days) and if pregnant up to 8 weeks after completion of cycle
  The primary endpoint of the trial is the Clinical Pregnancy Rate per cycle initiated

SECONDARY OUTCOMES:
Live birth rates | Up to 1 year or until delivery
  The secondary endpoint is the Live Birth Rate per cycle initiated (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel A Stadtmauer, MD, PhD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Laurel A. Stadtmauer, MD, PhD, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franks S. Assessment and management of anovulatory infertility in polycystic ovary syndrome. Endocrinol Metab Clin North Am. 2003 Sep;32(3):639-51. doi: 10.1016/s0889-8529(03)00044-6. PMID 14560891
- [Background] GOLDZIEHER JW, GREEN JA. The polycystic ovary. I. Clinical and histologic features. J Clin Endocrinol Metab. 1962 Mar;22:325-38. doi: 10.1210/jcem-22-3-325. No abstract available. PMID 13899931
- [Background] Richardson MR. Current perspectives in polycystic ovary syndrome. Am Fam Physician. 2003 Aug 15;68(4):697-704. PMID 12952386
- [Background] Hamilton-Fairley D, Taylor A. Anovulation. BMJ. 2003 Sep 6;327(7414):546-9. doi: 10.1136/bmj.327.7414.546. No abstract available. PMID 12958117
- [Background] Vendola KA, Zhou J, Adesanya OO, Weil SJ, Bondy CA. Androgens stimulate early stages of follicular growth in the primate ovary. J Clin Invest. 1998 Jun 15;101(12):2622-9. doi: 10.1172/JCI2081. PMID 9637695
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Ganesh A, Goswami SK, Chattopadhyay R, Chaudhury K, Chakravarty B. Comparison of letrozole with continuous gonadotropins and clomiphene-gonadotropin combination for ovulation induction in 1387 PCOS women after clomiphene citrate failure: a randomized prospective clinical trial. J Assist Reprod Genet. 2009 Jan;26(1):19-24. doi: 10.1007/s10815-008-9284-4. Epub 2009 Jan 7. PMID 19127427
- [Background] Casper RF. Aromatase inhibitors in ovarian stimulation. J Steroid Biochem Mol Biol. 2007 Aug-Sep;106(1-5):71-5. doi: 10.1016/j.jsbmb.2007.05.025. Epub 2007 May 24. PMID 17604615
- [Background] Eckmann KR, Kockler DR. Aromatase inhibitors for ovulation and pregnancy in polycystic ovary syndrome. Ann Pharmacother. 2009 Jul;43(7):1338-46. doi: 10.1345/aph.1M096. Epub 2009 Jul 7. PMID 19584394
- [Background] Miles RA, Paulson RJ, Lobo RA, Press MF, Dahmoush L, Sauer MV. Pharmacokinetics and endometrial tissue levels of progesterone after administration by intramuscular and vaginal routes: a comparative study. Fertil Steril. 1994 Sep;62(3):485-90. doi: 10.1016/s0015-0282(16)56935-0. PMID 8062942
- [Background] Cortinez A, De Carvalho I, Vantman D, Gabler F, Iniguez G, Vega M. Hormonal profile and endometrial morphology in letrozole-controlled ovarian hyperstimulation in ovulatory infertile patients. Fertil Steril. 2005 Jan;83(1):110-5. doi: 10.1016/j.fertnstert.2004.05.099. PMID 15652895
- [Background] Montville CP, Khabbaz M, Aubuchon M, Williams DB, Thomas MA. Luteal support with intravaginal progesterone increases clinical pregnancy rates in women with polycystic ovary syndrome using letrozole for ovulation induction. Fertil Steril. 2010 Jul;94(2):678-83. doi: 10.1016/j.fertnstert.2009.03.088. Epub 2009 Jun 9. PMID 19515366